CLINICAL TRIAL: NCT07313787
Title: Prospective Cross-Over Study of the Effects of Meal Macronutrients on Postprandial Lipids
Brief Title: Effects of Meal Macronutrients on Postprandial Lipids
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002465; 002465-DK
Record Dates: First submitted 2025-12-31; First posted 2026-01-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-16

CONDITIONS: Nephrotic Syndrome; Lipodystrophy; Metabolic Syndrome; Healthy Volunteer; Diabetes; Metabolic Associated Steatotic Liver Disease
Keywords: postprandial lipids; macronutrient; CARBOHYDRATES; FATS; Proteins
MeSH Terms: conditions — Nephrotic Syndrome; Lipodystrophy; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Healthy (Experimental): Healthy
  Interventions: Other: High carb then high fat breakfast; Other: High fat then high carb breakfast
- Lipodystrophy (Experimental): Lipodystrophy
  Interventions: Other: High carb then high fat breakfast; Other: High fat then high carb breakfast
- Metabolic syndrome (Experimental): Metabolic syndrome
  Interventions: Other: High carb then high fat breakfast; Other: High fat then high carb breakfast
- Nephrotic syndrome (Experimental): Nephrotic syndrome
  Interventions: Other: High carb then high fat breakfast; Other: High fat then high carb breakfast

INTERVENTIONS:
Other: High carb then high fat breakfast — High carb then high fat breakfast
Other: High fat then high carb breakfast — High fat then high carb breakfast

SUMMARY:
Background:

Abnormal fats in the blood can lead to many problems, including heart disease. Researchers want to learn more about how eating meals with different levels of nutrients affects fats in the blood. Specifically, they want to study people with too much body fat, too little body fat, and a kidney problem called nephrotic syndrome.

Objective:

To learn more about how different types of foods affect fat levels in the blood.

Eligibility:

People aged 18 years or older with a health condition that affects how their body handles fats. Healthy volunteers are also needed.

Design:

Participants will have 2 overnight stays in the clinic within 6 months. At each visit, after staying overnight, they will eat a breakfast casserole. At 1 visit, breakfast will be a high-fat, low carbohydrate meal. At the other, it will be a high-carbohydrate, low-fat meal.

Participants will have a tube inserted into a vein in their arm. They will have blood drawn via the tube 12 times in 8 hours: 2 times before they eat the breakfast and 10 times after.

Participants will have other tests during their stays:

* A resting metabolic test captures the air they exhale and measures how much energy they use at rest.
* A dual energy X-ray absorptiometry (DXA) scan measures how much fat and muscle they have.
* A Fibroscan is a special type of ultrasound of the liver.
* A body surface scan uses lasers to measure the total area of the body.
* A bioelectric impedance (BIS) exam measures how fast small electric currents move through their body.

Participants may opt to have a third visit. At this visit, the breakfast will be high in protein.

DETAILED DESCRIPTION:
Study Description:

This is a single site, randomized cross-over study assessing the effects of different test meals of varying macronutrient composition on post-prandial lipid metabolism. Studies will be conducted in healthy individuals and in several patient populations including those with nephrotic syndrome (NS), lipodystrophy, and metabolic syndrome.

The study hypothesis is that the number, composition and kinetics of lipid-containing particles will differ in the post-prandial state:

1. Within subjects, comparing meals of differing macronutrient composition (i.e. high fat versus high carbohydrate)
2. Between subjects with different disorders (i.e., lipodystrophy vs. NS vs. healthy)
3. Within subjects before and after treatment of their underlying disorders (i.e. nephrotic vs non-nephrotic states)

Objectives:

* Primary Objective: Determine the difference in postprandial triglycerides between meals of different macronutrient composition within each study cohort.
* Secondary Objective: Determine differences in post-prandial triglycerides between different study populations.

Endpoints:

* Primary Endpoint: Difference in baseline adjusted AUC for TG for 8 hours after meals of different macronutrient composition.
* Secondary Endpoints: Difference in baseline adjusted AUC for TG for each meal test between study cohorts

ELIGIBILITY:
* INCLUSION CRITERIA:

Common inclusion criteria (all groups):

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age >= 18 years
2. Average alcohol intake in the past 6 months < 30 g/day (male) or <20 g/day (female)

Healthy control specific inclusion criteria:

1. In good general health with no known active medical conditions as evidenced by medical history
2. Fasting glucose <100 mg/dL
3. HbA1c <5.7%
4. Fasting triglycerides <150 mg/dL
5. ALT and AST within normal limits
6. BMI >=18.5 to <25 kg/m^2 (or <23 kg/m^2 in participants of Asian descent)
7. Not taking any medications or supplements that, in the opinion of the investigator, would interfere with interpretation of study data.

Metabolic syndrome specific inclusion criteria

1. Obesity defined as either

1. BMI >30 kg/m^2 (or >=27 kg/m^2 in participants of Asian descent), OR
2. Elevated waist circumference as defined below:

   * Country/Ethnic group - Europid, Sub-Saharan African, Eastern Mediterranean and Middle East (Arab):

     --Sex: Male - Waist circumference: >=94cm

     --Sex: Female - Waist circumference: >=80cm
   * Country/Ethnic group - South Asian, Chinese, Japanese, Ethnic South and Central American:

     * Sex: Male - Waist circumference: >=90cm
     * Sex: Female - Waist circumference: >=80cm

       2. Elevated triglycerides defined as EITHER

       2a. Fasting triglycerides >= 150 mg/dL at screening, OR

       2b. Specific treatment for hypertriglyceridemia

       3. Low HDL cholesterol, defined as EITHER

       3a. HDL <40 mg/dL (males) or <50 mg/dL (females) at screening, OR

       3b. Specific treatment for low HDL

       4. Elevated blood pressure defined as EITHER

       4a. Systolic BP >= 130 at screening, OR

       4b. Diastolic BP >= 85 mm Hg at screening, OR

       4c. Treatment of previously diagnosed hypertension

       5. Elevated glucose defined as EITHER

       5a. HbA1c >= 5.7% (at screening), OR

       5b. Fasting serum glucose >= 100 mg/dL (at screening), OR

       5c. 2-hour post-load glucose levels >= 140 mg/dL (by history), OR

       5d. Prior diagnosis of type 2 diabetes

   Lipodystrophy-specific inclusion criteria:
   1. Clinical diagnosis of generalized or partial lipodystrophy based on reduction in adipose tissue outside the normal range in some or all adipose depots (including, at aminimum, the gluteofemoral depot).
   2. Insulin resistance as defined by fasting insulin >22.5 or high exogenous insulin requirement (> 2 units per kg per day or > 200 units total per day) at screening.

   Nephrotic syndrome specific inclusion criteria
   1. History of biopsy proven non-diabetic glomerular disease (any histology)
   2. Nephrotic range proteinuria defined by ANY of the following:

   2a. Protein/creatinine ratio uPCR >= 3.5 g/g at screening, OR

   2b. 24 hour protein excretion >= 3.5 gr/24hr) at screening, OR

   2c. History of nephrotic range proteinuria (as defined above) within the past 5 years but in complete (defined as proteinuria <= 0.3 g/day or partial remission (defined as a 50% or greater decrease in proteinuria compared to baseline and proteinuria < 3.5 g/day) based on 24 hr urine or uPCR at time of screening

   EXCLUSION CRITERIA:

   Common exclusion criteria (all groups):

   An individual who meets any of the following criteria will be excluded from participation in this study:
   1. Consuming extreme macronutrient diet (e.g., very low-carbohydrate, high fat diets such as ketogenic, paleo or Atkins diets, among others).
   2. Plans to actively gain or lose weight during the study period (other than changes in water balance as clinically needed in subjects with nephrotic syndrome).
   3. Change in body weight of >5% or >3 kg (whichever is larger) in the 3 months prior to screening (by participant report) in participants who do NOT have nephrotic syndrome.
   4. Body weight >450 lbs (upper limit that can be accommodated by DXA scanner).
   5. Participating in a regular strenuous exercise program (> 2h/week of vigorous activity) as determined by volunteer report or evidence of vigorous exercising in order to lose weight, change body shape, or to counteract the effects of eating.
   6. Uncontrolled diabetes, defined as HbA1c >9% at screening.
   7. Lipemia defined as fasting or non-fasting triglycerides of >1000 mg/dL at screening.
   8. Renal dysfunction defined as eGFR <50 mL/min/1.73 m^2 at screening.
   9. In participants with liver disease, history of decompensated advanced liver disease, defined as direct bilirubin > 0.5 g/dL, PT > 18 seconds, albumin < 3 g/dL, MELD score > 12, or history of ascites, encephalopathy, variceal bleeding, spontaneous bacterial

      peritonitis or liver transplant.
   10. History of hypertriglyceridemia-induced pancreatitis within 3 months prior to screening.
   11. Positive pregnancy test or breastfeeding at screening.
   12. Clinically significant abnormalities in thyroid function, blood counts, as assessed by screening labs.
   13. Acute cardiovascular events within the past 6 months
   14. Anemia (Hgb <10 mg/dL in women or <12 mg/dL in men) at screening
   15. Food allergies or other dietary restrictions that could increase risk associated with test meals or cause the subject to be unwilling to consume test meals (i.e. celiac disease, vegan diets).
   16. Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, or other known conditions that could affect intestinal fat absorption.
   17. Subjects treated with tamoxifen, estrogens, or progestins that have not been stable for >4 weeks prior to screening.
   18. Blood donation in the last 2 weeks or planned blood donation during the study
   19. Subjects requiring regular transfusions for any reason.
   20. Subjects with known gastroparesis
   21. Inability to adhere to Lifestyle Considerations throughout study duration.
   22. Inability of the subject to understand and the unwillingness to sign a written informed consent document.
   23. Unwillingness to comply with all study procedures and unavailable for the duration of the study
   24. Any other condition or medication which, in the opinion of the investigator, increases risk to the subject, prevents the subject from complying with study procedures, prevents the subject from completing the study, or interferes with the interpretation of study results.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Determine the difference in postprandial triglycerides between meals of different macronutrient composition within each study cohort. | 8 hours
  Difference in baseline adjusted AUC for TG for 8 hours after meals of different macronutrient composition.

SECONDARY OUTCOMES:
Determine differences in post-prandial triglycerides between different study populations. | 8 hours
  Difference in AUC for TG for each meal test between study cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will collect data from subjects enrolled at the NIH Clinical Center to meet the primary and secondary endpoints as stated in the protocol. Demographic, laboratory results, clinical observations and imaging studies will be acquired from up to 100 participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Scientific data included in published manuscripts will be made available at the time of publication; all other generated scientific data will be shared no later than the termination date of the study. The study data will be stored in the repository for at least 5 years.
Access Criteria: Identifiable data will be de-identified prior to repository submission. Participant-level clinical data described above will be preserved through deposition of the data in a controlled access public repository. Scientific data included in published manuscripts will be made available at the time of publication; all other generated scientific data will be shared no later than the termination date of the study.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002465-DK.html